CLINICAL TRIAL: NCT00081159
Title: A Randomized Phase II Study Of Bone-Targeted Therapy In Advanced Androgen-Dependent Prostate Cancer
Brief Title: Hormone Ablation Therapy, Doxorubicin, and Zoledronate With or Without Strontium 89 in Treating Patients With Androgen-Dependent Prostate Cancer and Bone Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0922; MDA-2003-0922; NCI-6459; NCI-2009-00062 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); CDR0000360625 (Other: NCI); 2U10CA045809-17 (NIH)
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Results first posted 2016-11-10 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-09

CONDITIONS: Metastatic Cancer; Prostate Cancer
Keywords: recurrent prostate cancer; stage IV prostate cancer; bone metastases
MeSH Terms: conditions — Neoplasm Metastasis; Prostatic Neoplasms | interventions — Doxorubicin; Goserelin; Leuprolide; Zoledronic Acid; Orchiectomy; strontium chloride; Strontium-89

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HAT, Doxorubicin, Zoledronate + Strontium chloride (Experimental): Arm I: Hormonal ablative therapy (HAT) comprising luteinizing hormone-releasing hormone agonist (e.g., leuprolide or goserelin) continuously during study treatment OR bilateral orchiectomy; doxorubicin IV on days 1, 8, and 15 every 28 days for 2 courses; zoledronate IV over 15 minutes on day 1 every 28 days for 6 courses; and a single dose of strontium chloride Sr 89 IV over 1-2 minutes on day 1.
  Interventions: Drug: Doxorubicin hydrochloride; Drug: Goserelin acetate; Drug: Leuprolide acetate; Drug: Zoledronic acid; Procedure: orchiectomy; Radiation: strontium chloride Sr
- HAT, Doxorubicin + Zoledronate (Experimental): Arm II: HAT, doxorubicin, and zoledronate as in arm I. HAT comprising luteinizing hormone-releasing hormone agonist (e.g., leuprolide or goserelin) continuously during study treatment OR bilateral orchiectomy; doxorubicin IV on days 1, 8, and 15 every 28 days for 2 courses; zoledronate IV over 15 minutes on day 1 every 28 days for 6 courses.
  Interventions: Drug: Doxorubicin hydrochloride; Drug: Goserelin acetate; Drug: Leuprolide acetate; Drug: Zoledronic acid; Procedure: orchiectomy

INTERVENTIONS:
Drug: Doxorubicin hydrochloride — Doxorubicin 20 mg/m^2 is administered intravenously either over 15 to 30 minutes via a peripheral line or over 24 hours via a central line on days 1, 8, and 15 every 28 days for 2 cycles.
  Other Names: Adriamycin PFS; Adriamycin RDF; Adriamycin; Rubex
Drug: Goserelin acetate
  Other Names: Zoladex
Drug: Leuprolide acetate
  Other Names: Lupron Depot
Drug: Zoledronic acid — 4 mg given intravenously over 15 minutes every 28 days for a total of 6 doses.
  Other Names: Zoledronate; Zometa
Procedure: orchiectomy
Radiation: strontium chloride Sr — 1 dose of strontium-89 (4 millicurie (mCi) total dose) administered intravenously on the first day of treatment
  Other Names: Sr-89; Strontium-89; Mestastron
  Arms: HAT, Doxorubicin, Zoledronate + Strontium chloride

SUMMARY:
RATIONALE: Androgens can stimulate the growth of prostate cancer cells. Drugs such as goserelin and leuprolide may fight prostate cancer by stopping the adrenal glands from producing androgens. Drugs used in chemotherapy such as doxorubicin work in different ways to stop tumor cells from dividing so they stop growing or die. Zoledronate may prevent bone loss and stop the growth of tumor cells in bone. Radioactive substances such as strontium-89 may relieve bone pain associated with prostate cancer. It is not yet known whether hormone (androgen) ablation therapy and chemotherapy combined with zoledronate is more effective with or without strontium-89 in treating prostate cancer and bone metastases.

PURPOSE: This randomized phase II trial is studying giving hormone ablation therapy, doxorubicin, and zoledronate together with strontium-89 to see how well it works compared to hormone ablation therapy, doxorubicin, and zoledronate alone in treating patients with androgen-dependent prostate cancer and bone metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the clinical efficacy of hormonal ablative therapy combined with doxorubicin and zoledronate with or without strontium chloride Sr 89, in terms of progression-free survival, in patients with androgen-dependent prostate cancer and bone metastases.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to the number of bony metastases (≤ 6 versus > 6). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive hormonal ablative therapy comprising luteinizing hormone-releasing hormone agonist (e.g., leuprolide or goserelin) continuously during study treatment OR bilateral orchiectomy. Patients also receive doxorubicin intravenously (IV) on days 1, 8, and 15 every 28 days for 2 courses; zoledronate IV over 15 minutes on day 1 every 28 days for 6 courses; and a single dose of strontium chloride Sr 89 IV over 1-2 minutes on day 1.
* Arm II: Patients receive hormonal ablative therapy, doxorubicin, and zoledronate as in arm I.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 80 patients (40 per treatment arm) will be accrued for this study within 20 months.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed prostate carcinoma.
2. Osteoblastic metastases on bone scan or computed tomography (CT) scan.
3. Initiation of hormonal ablative therapy within 3 months of registration.
4. Prior neoadjuvant, concurrent, or intermittent hormonal ablative therapy of less than 3 years duration and completed at least 3 years prior to entry into this study.
5. The Eastern Cooperative Oncology Group (ECOG) performance status <3 (Karnofsky >40%)
6. Patients must have normal organ and marrow function as defined: leukocytes: >3,000/mL; absolute neutrophil count: >1,500/mL; platelets: >100,000/mL; total bilirubin within normal institutional limits; alanine transaminase (ALT)(SGPT)/aspartate aminotransferase (AST)(SGOT): <2.5 * institutional upper limit of normal; creatinine: < or = 3.0; left ventricular ejection fraction: >45%
7. The effects of strontium-89 and zoledronic acid on the developing human fetus at the recommended therapeutic dose are unknown. Even though all patients are castrated during this study, men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should the spouse of a patient become pregnant or suspect she is pregnant while participating in this study, she/he should inform the treating physician immediately.
8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. More than one prior chemotherapy regimen. Prior doxorubicin treatment is permitted. However patient's with >250 mg/m2 cumulative dosage are excluded.
2. Prior radioisotope treatment consisting of strontium-89 or samarium-153.
3. Zoledronic acid treatment for more than 3 months duration prior to registration. Other bisphosphonate treatments are permitted.
4. Corrected serum calcium level less than 8 mg/dL.
5. Patients may not be receiving any other investigational agents.
6. Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to zoledronic acid or other agents used in the study
8. Patients with the following atypical presentations should have a biopsy: those with small cell carcinoma, purely lytic bone metastases, or bulky (i.e. 5 cm) visceral or nodal disease in the absence of bone involvement are not eligible.
9. Symptomatic bulky lymphadenopathy causing scrotal or pedal edema or significant local invasive disease in bladder invasion.
10. History of other malignancies other than nonmelanoma skin cancer, unless in complete remission and off therapy for that disease for at least 5 years.
11. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, history of congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
12. Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with strontium-89 or other agents administered during the study. Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.
13. Evidence or suspicion of myelodysplastic syndrome by complete blood test (CBC) must be confirmed by bone marrow biopsy.
14. Untreated symptomatic spinal cord compressions.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Ming Tu, MD, Study Chair — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - CCOP - Wichita, Wichita, Kansas
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: July 6, 2004 to July 5, 2007. Recruitment done in medical clinic settings.
Pre-assignment Details: One participant of 80 male participants withdrew consent after the screening procedures therefore was not randomized nor treated and is excluded from the trial.
Groups:
- HAT, Doxorubicin, Zoledronate + Strontium Chloride: Arm I: Hormonal ablative therapy (HAT) comprising luteinizing hormone-releasing hormone agonist (e.g., leuprolide or goserelin) continuously during study treatment OR bilateral orchiectomy; doxorubicin intravenous (IV) on days 1, 8, and 15 every 28 days for 2 courses; zoledronate IV over 15 minutes on day 1 every 28 days for 6 courses; and a single dose of strontium chloride Sr 89 IV over 1-2 minutes on day 1.
Period: Overall Study
Arm/Group | HAT, Doxorubicin, Zoledronate + Strontium Chloride | HAT, Doxorubicin + Zoledronate
Started | 39 | 40
Completed | 37 | 35
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Myelosuppression prior to treatment | 0 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HAT, Doxorubicin, Zoledronate + Strontium Chloride | HAT, Doxorubicin + Zoledronate | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Continuous [Median (Full Range); unit: years] | 62 [46 to 77] | 63 [46 to 82] | 63 [46 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 39 | 40 | 79
Race/Ethnicity, Customized [Number; unit: participants]
  White | 37 | 34 | 71
  Black | 2 | 3 | 5
  Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 39 | 40 | 79

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Study's primary endpoint of PFS duration/time to progression was defined as the time from the date of randomization to the date of first evidence of disease progression or patient death. Prostate-specific antigen (PSA) progression is usually the first evidence of progression. PSA progression is defined as a 25% increase over the baseline or the nadir provided that the increase is a minimum of 1 ng/ml.
Time Frame: Up to 90 months with evaulation in 4 week intervals for up to 6 months of treatment, then follow up until disease progression
Population: Intent to treat population analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HAT, Doxorubicin, Zoledronate + Strontium Chloride | HAT, Doxorubicin + Zoledronate
Number analyzed (Participants) | 39 | 40
Months | 12.9 [8.9 to 72.5] | 18.5 [9.7 to 49.4]

2. Secondary Outcome: Major Bone Scan Response
Description: Bone scan performed at baseline and at Week 13 provided if baseline scan was positive for metastases. A major bone scan response was considered with a substantial resolution of participant bone metastases on the bone scans, i.e. complete resolution of the osseous metastases on the bone scan.
Time Frame: Week 13
Population: Five participants in the non-Strontium arm were not evaluable for this outcome, four withdrew prior to treatment, and one had disease progression that precluded inclusion. Two participants in the Strontium arm were lost to follow up therefore excluded from analysis as well.
Measure: Number; unit: participants
Arm/Group | HAT, Doxorubicin, Zoledronate + Strontium Chloride | HAT, Doxorubicin + Zoledronate
Number analyzed (Participants) | 37 | 35
participants | 0 | 0

3. Other Pre Specified Outcome: Overall Survival (OS)
Description: Overall Survival defined as the length of time from the start of treatment till time that participants are still alive.
Time Frame: Up to 90 months
Population: Intent to treat population analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HAT, Doxorubicin, Zoledronate + Strontium Chloride | HAT, Doxorubicin + Zoledronate
Number analyzed (Participants) | 39 | 40
Months | 47.4 [35.9 to 87.3] | 53.5 [38.0 to NA] — Not attainable, time constraint

ADVERSE EVENTS:
Time Frame: Adverse event collection from beginning of treatment through week 21, and up to week 24 post treatment.
Description: Three of the 40 participants in the Non-Strontium arm (Arm 2) did not receive treatment and are therefore excluded from Adverse Event reporting.
Arm/Group | HAT, Doxorubicin, Zoledronate + Strontium Chloride | HAT, Doxorubicin + Zoledronate
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/37
Other Adverse Events (participants affected / at risk) | 24/39 | 29/37
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HAT, Doxorubicin, Zoledronate + Strontium Chloride (N=39) | HAT, Doxorubicin + Zoledronate (N=37)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Alt, Sgpt) (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Ast, Sgot) (Investigations) | 0 (0) | 1 (1)
Bilirubin Increased (Investigations) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 5 (5) | 6 (6)
Fever Without Neutropenia (General disorders) | 0 (0) | 3 (3)
Flu-Like Syndrome (General disorders) | 1 (1) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hemoglobin Increased (Investigations) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Mood Alteration (Psychiatric disorders) | 1 (1) | 0 (0)
Mucositis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (5)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0)
Pain (Back) (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain (Extremity-Limbs) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain (Face) (General disorders) | 1 (1) | 0 (0)
Pain (Joint) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes